CLINICAL TRIAL: NCT02827851
Title: Evaluation of Safety and Effectiveness of Intraarticular Administration of Autologous Stromal Vascular Fraction of Cells for Treatment of Knee Articular Cartilage Dystrophy
Brief Title: Autologous Stromal Vascular Fraction of Cells for Treatment of Knee Articular Cartilage Dystrophy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Collaborators: Orenburg Regional Clinical Blood Donor Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-ССН-03-01-16
Record Dates: First submitted 2016-06-24; First posted 2016-07-11 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Knee Osteoarthritis
Keywords: Damage of articular cartilage; Cartilage degeneration; Intraarticular injection; SVF; Stromal vascular fraction; Adipose-derived regenerative cells (ADRC); Adipose tissue; Stem cells
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SVF injection (Experimental): Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate stromal vascular fraction of cells (SVF). After SVF isolation autologous cells suspension will be injected intraarticularly into knee joint.
  Interventions: Procedure: Liposuction; Other: SVF isolation; Other: Intraarticular administration of autologous SVF

INTERVENTIONS:
Procedure: Liposuction
Other: SVF isolation — SVF will be isolated according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 5 ml of Hartmann's solution.
Other: Intraarticular administration of autologous SVF

SUMMARY:
Stromal vascular fraction of cells (SVF) will be extracted from lipoaspirate by enzymatic digestion. SVF will be administered in a single dose intraarticularly 4 weeks after arthroscopic debridement. All patients will receive cell therapy.This is a single arm study with no control.

DETAILED DESCRIPTION:
Patients undergone arthroscopic debridement for knee osteoarthritis will be subjected to abdominal liposuction under local anaesthesia. Harvested adipose tissue will be processed according to patent pending technology based on enzymatic digestion, washing and concentration of cell pellet in 5 ml of Hartmann's solution. Isolated SVF will be administered in a single dose into anterior part of knee joint cavity 28 days after arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the knee joint during more than a half day assessed by Visual Analog Pain Scale (score more than 40 mm)
* At least three of the following 6 criteria: 50 years of age or older, stiffness lasting less than 30 minutes, crepitus, bony tenderness, bony enlargement, no warmth to the touch
* Patient is able to walk without assistance
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Medical history of endoprosthetic knee replacement
* Medical history of lower extremity osteotomy
* Medical history of knee surgery (including arthroscopy) during preceding 1 year prior to enrollment
* Medical history of intraarticular injections during preceding 6 months prior to enrollment
* Secondary osteoarthritis of the knee joint: posttraumatic osteoarthritis (developed after clinically significant injury), intra-articular fractures, clinically significant varus or valgus deformities of lower limbs, septic arthritis, joint's inflammatory disorders, gout, advanced chondrocalcinosis, Paget's disease, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary synovial osteochondromatosis, osteonecrosis, hemophilia
* Patients prescribed for immunosuppressive treatment
* Medical history of systemic autoimmune and inflammatory diseases
* Significant weight loss (> 10% of body weight in the previous year) of unknown etiology
* Medical history of venous thromboembolism or estimated high risk of venous thromboembolism
* Patients prescribed for systemic corticosteroids or other medications treatment with proven impact on bone or cartilage tissue metabolism
* Clinically significant abnormalities in results of laboratory tests
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy.
* Patient's activated partial thromboplastin time exceeds normal levels more than 1,8 times
* Patients prescribed for anticoagulants treatment or patient received anticoagulants at least one hour prior liposuction
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Patient's refusal from compliance with the requirements of contraception during the participation in research
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockcroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

* Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
SAEs monitoring | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse events (SAEs)
SARs monitoring | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse reactions (SARs)

SECONDARY OUTCOMES:
Quality of life monitoring-1 | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaire - the Short Form (36) Health Survey (SF-36)
Quality of life monitoring-2 | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaire - Knee Injury and Osteoarthritis Outcome Score (KOOS)
Knee pain intensity monitoring | Follow up to completion (up to 24 weeks after treatment)
  Knee pain intensity assessed by Visual Analog Pain Scale (no pain=0; maximum pain=100 mm)
Changes in knee joint structure-1 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by ultrasonography (effusion, synovial thickening or hypertrophy, cartilage parameters, vascularity, Baker's cysts, osteophytes, tendon and ligament abnormalities, meniscal changes, bursitis, erosions and panniculitis)
Changes in knee joint structure-2 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by X-ray (joint space width, bone contour, presence of osteophytes and sclerosis)
Changes in knee joint structure-3 | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by MRI (articular cartilage, osteophytes, bone marrow abnormality, meniscal integrity, synovial effusion/tissue, anterior and posterior cruciate ligaments, and medial and lateral collateral ligaments)
Changes in knee function | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee function assessed by validated questionnaire: Knee Society Score (KSS)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya I Eremin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies; Rinat G Gilmutdinov, MD, PhD, Principal Investigator — Orenburg Regional Clinical Donor Blood Center; Sergey I Gilfanov, MD, PhD, Prof, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Andrey A Averyanov, MD, PhD, Principal Investigator — Orenburg Regional Clinical Hospital; Vadim A Kopylov, MD, PhD, Principal Investigator — Orenburg City Clinical Hospital #4
Locations (4):
- Russia (4):
  - Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation, Moscow
  - Orenburg City Clinical Hospital #4, Orenburg
  - Orenburg Regional Clinical Donor Blood Center, Orenburg
  - Orenburg Regional Clinical Hospital, Orenburg

IPD SHARING:
Plan to Share IPD: Undecided